CLINICAL TRIAL: NCT02874482
Title: Study of Cognitive and Emotional Factors Influencing the Visual Exploration Among Patients With Schizophrenia
Brief Title: Cognitive and Emotional Factors in Visual Exploration Among Patients With Schizophrenia
Acronym: SAILLANCE1
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_19.1; 2013-A01497-38 (Other: ANSM)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Change blindness; Eye tracking; Implicit response
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with schizophrenia: 30 patients with schizophrenia (diagnosis based on the standard DSM criteria)
- Controls: 30 healthy controls without any psychiatric or neurological diagnosis

SUMMARY:
Background:

Patients with schizophrenia are abnormally disturbed by information onsets, which may result in a disadvantage in filtering relevant information. It seems that they accord the same importance to all objects in a scene without taking into account the relevance of objects (cognitive salience) or their emotional charge (salience emotional).

The paradigm of change blindness offers the interesting possibility of studying sensitivity to the sudden irruption of visual information with ecological stimuli in schizophrenia. An increased attentional capture by the irruption of visual information would suggest better performance in patients than in healthy controls. Moreover, patients are disturbed to processing of emotional information, in this way we would like to measure the impact of emotional salience on the visual exploration.

Main aim:

The main objective is to evaluate, if patients with schizophrenia quickly detect changes occurring on irrelevant objects in the understanding of the scene.

Secondary objectives:

To evaluate in patients with schizophrenia the impact of emotional salience using the same paradigm.

To separate an explicit response (motors responses) with an implicit response (eye tracking measures).

Methodology:

30 patients with schizophrenia and 30 healthy controls were asked to detect changes in 96 scenes with 0 or 1 change (neutral or emotional changes). We will measure the participants' speed and accuracy in explicitly reporting the changes via motor responses and their capacity to implicitly detect changes via eye movements.

DETAILED DESCRIPTION:
This study will include one visit:

* Written consent will be obtained from all participants
* Inclusion and exclusion criteria will be checked
* An ophthalmologic test, a pregnancy test, a alcohol test and a salivary test will be realized
* Various symptoms will be assessed with the PANSS (Positive And Negative Syndrome Scale for schizophrenia) and the UPDRS (Unified Parkinson Disease Rating Scale for patients, the MOCA (Montreal Cognitive Assessment), The HAD (Hospital Anxiety and Depression Scale) and the MINI (Mini International Neuropsychiatric Interview) for all participants.
* The task will be divided in two parts:

A visuo-spatial task allowing to record saccadic eye movements (approximately 10 min).

The change blindness session lasted approximately 20 min.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected vision
* Affiliate to a social security system
* For group of patients with schizophrenia : diagnosis of schizophrenia based on the standard DSM-IV criteria and patients will be clinically stable at the testing time

Exclusion Criteria:

* History of neurological illness
* Pregnant and nursing women
* Drugs use in the last 24 hours
* Acute ocular disorder
* Under tutorship, curatorship or deprived of liberty
* For controls group : be free DSM-IV axis-I diagnoses according the MINI test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients with schizophrenia and 30 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-11-17 (Actual); Study Completion 2019-11-17 (Actual)

PRIMARY OUTCOMES:
response time | 42 months
  The explicit response of the participants will be measure behaviourally by response time before the detection of neutral stimuli.

SECONDARY OUTCOMES:
sensitivity index | 42 months
  Performances will be measure by a sensitivity index (D prime) which considers the number of correct detections compared with the missed detections and false alarms; thus it evaluates the capacity to discriminate the signal against a background noise.
implicit response | 42 months
  The implicit response will be measure by the localization and duration of fixations
emotional response | 42 months
  The emotional response will be measure by the localization, duration of fixations and performances for the detection of emotional stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume VAIVA, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital, Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No